CLINICAL TRIAL: NCT05880160
Title: Randomised Control Trial for the Safety of Withdrawal of Pharmacological Treatment for Recovered HER2 Targeted Therapy Related Cardiac Dysfunction
Brief Title: Safety of Withdrawal of Pharmacological Treatment for Recovered HER2 Targeted Therapy Related Cardiac Dysfunction
Acronym: HER-SAFE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Collaborators: British Heart Foundation (Other); Barts & The London NHS Trust (Other); University College London Hospitals (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 147133; FS/CRTF/22/24395 (Other Grant/Funding Number: British Heart Foundation); 312432 (Other: IRAS)
Record Dates: First submitted 2023-02-08; First posted 2023-05-30 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Cardiotoxicity; HER2-positive Breast Cancer; Heart Failure; Cancer, Therapy-Related
Keywords: Cardiotoxicity; HER2-positive Breast Cancer; Heart Failure; Cancer, Therapy-Related
MeSH Terms: conditions — Cardiotoxicity; Heart Failure; Neoplasms, Second Primary

STUDY DESIGN:
Intervention Model Description: Two centre open label randomised control trial to evaluate the phased withdrawal versus continuation of heart failure treatment for 'recovered' human epidermal growth factor receptor 2 (HER2) therapy-related cardiac dysfunction in non-high risk patients following completion of HER2 therapy.
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Withdrawal (Experimental): Participants will undergo phased withdrawal of heart failure/ cardioprotective treatments according to a pre-specified algorithm based on the 'Withdrawal of pharmacological treatment for heart failure in patients with recovered dilated cardiomyopathy' (TRED-HF) study protocol (Halliday et al 2019). Medications will be down titrated in a phased process every 2 weeks over 16 weeks maximum. Drug doses will be reduced by 50% every 2 weeks, until the patient is taking 25% or less of the maximum recommended dose at which point they will be stopped. Monitoring with fortnightly virtual consultations will confirm dose reduction and provide support. Participants will undergo clinical assessment at 6, 14 and 24 weeks and 6, 9 and 12 months with weight, blood pressure, and biomarker measurement. At baseline, 6- and 12-month visits detailed cardiovascular phenotyping using cardiovascular magnetic resonance scans and symptom and disutility questionnaires will be undertaken.
  Interventions: Other: Phased withdrawal of heart failure medications
- Treatment Continuation (No Intervention): Participants will continue their current heart failure/ cardioprotective treatments. Participants will undergo clinical assessment at 6, 14 and 24 weeks and 6, 9 and 12 months with weight, blood pressure, and biomarker measurement. At baseline, 6- and 12-month visits detailed cardiovascular phenotyping using cardiovascular magnetic resonance scans and symptom and disutility questionnaires will be undertaken.

INTERVENTIONS:
Other: Phased withdrawal of heart failure medications — As per arm/group description
  Arms: Treatment Withdrawal

SUMMARY:
Breast cancer is the most common cancer in the United Kingdom (UK), but improvements in treatment mean 3 in 4 people survive for more than 10 years. Many people receive treatments called human epidermal growth factor receptor 2 (HER2) targeted therapies for their breast cancer, however these can affect heart function. This 'cardiotoxicity' is generally temporary and mild, but patients receive drugs to help their heart recover. Currently it is not known how long patients should receive these treatments. Patients with other types of heart failure are treated lifelong, but this may not be necessary here as the damaging cancer drugs have stopped. Taking drugs for many years can have an impact on people's quality of life, particularly for young patients. It is therefore important to understand the best treatment length. The investigators will study people whose heart function has recovered after HER2 therapy heart problems and are not at high risk for heart disease. The investigators will carefully stop their heart drugs whilst monitoring them closely with special heart scans and blood tests to detect problems early. The investigators will also study how patients are currently treated using national data. The results of this study will help doctors better guide breast cancer survivors about treatment of heart damage from HER2 cancer therapies.

DETAILED DESCRIPTION:
Trial design: Two centre open label randomised control trial to evaluate the phased withdrawal versus continuation of heart failure treatment for 'recovered' human epidermal growth factor receptor 2 (HER2) therapy-related cardiac dysfunction in non-high risk patients following completion of HER2 therapy. The trial will include cardiovascular magnetic resonance scans (CMR) with automated in-line analytics to improve the sensitivity for detection of early relapse, and detailed patient questionnaires assessing medication disutility to better understand participant motivations and concerns related to treatment continuation and withdrawal.

Trial population: The trial will recruit 90 adult participants (>18 years) with a prior diagnosis of HER2-targeted therapy related cardiac dysfunction, who currently receive standard heart failure/ cardioprotective medications (any combination of Angiotensin-converting enzyme [ACE] inhibitors, angiotensin receptor blockers [ARBs] and/or beta-blockers), and whose cardiac function has 'recovered'. 'Recovery' is defined as absence of heart failure symptoms with left ventricular ejection fraction (LVEF) improved to 50% or greater and N-terminal pro B-type natriuretic peptide (NTproBNP) <200ng/L, for greater than 6 months. Patients will be recruited from Barts Health and University College London Hospitals (UCLH) cardio-oncology and breast cancer clinics. Exclusion criteria: Patients with advanced/ metastatic HER2 positive breast cancer requiring ongoing HER2 therapies or with life expectancy <12months will be excluded. Patients classed as high/very high cardiotoxicity risk according to the European Society of Cardiology/International Cardio-Oncology Society Position Statement (Lyon et al, 2020), LVEF <50% prior to HER2-therapies or on completion of anthracycline treatment, or indications for ongoing ACE inhibitors, ARBs and/or beta-blockers, nor those with absolute contraindications to CMR.

Interventions and Duration of treatment: Participants will undergo phased withdrawal of heart failure/ cardioprotective treatments according to a pre-specified algorithm based on the 'Withdrawal of pharmacological treatment for heart failure in patients with recovered dilated cardiomyopathy' (TRED-HF) study protocol (Halliday et al 2019). This had been designed following extensive consultation with independent experts and attempts to mimic 'real-world' medication withdrawal in clinical practice. Medications will be down titrated in a phased process every 2 weeks over a maximum of 16 weeks. Drug doses will be reduced by 50% in a stepwise manner every 2 weeks, until the patient is taking 25% or less of the maximum recommended dose at which point the medication will be stopped. Monitoring with fortnightly virtual consultations will confirm drug dose reduction and provide support. Participants will undergo clinical assessment at 6, 14 and 24 weeks and 6, 9 and 12 months with weight, blood pressure, and biomarker measurement. At baseline, 6- and 12-month visits detailed cardiovascular phenotyping using CMR and symptom and disutility questionnaires will be undertaken.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants (>18 years)
2. A prior diagnosis of human epidermal growth factor receptor 2 (HER2)- targeted therapy related cardiac dysfunction, who currently receive standard heart failure/cardioprotective medications (any combination of angiotensin-converting enzyme [ACE] inhibitors, angiotensin receptor blockers [ARBs] and/or beta-blockers).
3. Cardiac function has 'recovered'. 'Recovery' is defined as absence of heart failure symptoms with left ventricular ejection fraction (LVEF) improved to 50% or greater and N-terminal pro B-type natriuretic peptide (NTproBNP) <125ng/L, for greater than 6 months.

Exclusion Criteria:

1. Advanced/ metastatic HER2 positive breast cancer requiring ongoing HER2 therapies or with life expectancy <12months.
2. Patients classed as high/very high cardiovascular risk according to the International Cardio-Oncology Society (ICOS) risk stratification
3. Patients with LVEF <50% prior to HER2-therapy initiation or on completion of anthracycline treatment
4. Patients with ongoing indications for the cardioprotective medication - ACE inhibitors, ARBs and/or beta-blockers
5. Patients with absolute contraindications to cardiovascular magnetic resonance scans (CMR).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Relapse in Cardiotoxicity | 12 months
  Number of participants with relapse in cardiotoxicity, defined based on International Cardio-Oncology Society 2021 Guidelines as (at least one of):
  1. Asymptomatic left ventricular ejection fraction (LVEF) reduction by ≥10 percentage points to a LVEF of <50%
  2. Asymptomatic LVEF reduction by ≥5 percentage points to an LVEF of <50% plus new relative decline in global longitudinal strain (GLS) by >15% from baseline AND/OR new rise in cardiac biomarkers (>2 fold increase in N-terminal pro B-type natriuretic peptide [NTproBNP] to >400ng/L, or high sensitivity Troponin >99th percentile)
  3. Clinical heart failure (based on symptoms and clinical examination) with at least one of the following: fall in LVEF ≥5%, increase in cardiac biomarkers (as above), relative fall in GLS > 15%, new arrhythmia (excluding ectopy)

SECONDARY OUTCOMES:
Cardiac Biomarkers (N-terminal pro B-type natriuretic peptide [NT-proBNP]) | 12 months
  Change from baseline at 6 and 12 months in the cardiac biomarker NT-proBNP (measured in pg/L)
Cardiac Biomarkers (Troponin T) | 12 months
  Change from baseline at 6 and 12 months in the cardiac biomarkers Troponin T (measured in ng/L).
Quality of life (Kansas City Cardiomyopathy Questionnaire) | 12 months
  Change from baseline at 6 and 12 months in the quality of life questionnaire score - the Kansas City Cardiomyopathy Questionnaire (Minimum 0 - Maximum 100; 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent).
Quality of life (Minnesota Living with Heart Failure Questionnaire) | 12 months
  Change from baseline at 6 and 12 months in quality of life questionnaire score - the Minnesota Living with Heart Failure Questionnaire (Minimum 0 - Maximum 105, Higher score indicates worse outcome).
Heart rate | 12 months
  Change from baseline at 6 and 12 months in baseline resting heart rate (beats per minute)
Blood Pressure | 12 months
  Change from baseline at 6 and 12 months in blood pressure (Systolic and diastolic, mmHg)
Left Ventricular Volumes (By Cardiac MRI) | 12 months
  Change from baseline at 6 and 12 months in CMR-derived left ventricular volumes (measured in ml and ml/m2)
Left Ventricular Ejection Fraction (By Cardiac MRI) | 12 months
  Change from baseline at 6 and 12 months in CMR-derived left ventricular ejection fraction (measured in %)
Left Ventricular Strain (By Cardiac MRI) | 12 months
  Change from baseline at 6 and 12 months in CMR-derived left ventricular strain (measured in %)
T1 mapping (By Cardiac MRI) | 12 months
  Change from baseline at 6 and 12 months in CMR-derived native T1 mapping (measured in ms)
Medication Disutility | 12 months
  Medication disutility is the inconvenience to the patient of taking a given medication. This will be assessed with a structured questionnaire with qualitative responses regarding medication side effects, cost (financial and personal) and the benefits required to offset this.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Manisty, Principal Investigator — UCL
Locations (2):
- United Kingdom (2):
  - St Bartholemew's Hospital, London
  - University College London Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dowsing B, Dehbi HM, Chung R, Pedra J, Worn O, Artico J, Schmid P, Roylance R, Kellman P, Moon JC, Crake T, Westwood M, Ghosh A, Andres MS, Nazir MS, Lyon AR, Chen D, Walker M, Manisty CH. HER-SAFE study design: an open-label, randomised controlled trial to investigate the safety of withdrawal of pharmacological treatment for recovered HER2-targeted therapy-related cardiac dysfunction. BMJ Open. 2025 Feb 5;15(2):e091917. doi: 10.1136/bmjopen-2024-091917. PMID 39909533